CLINICAL TRIAL: NCT06000254
Title: Efficacy of High Energy Density Pulse Electromagnetic Field for Patients With Adhensive Capsulitis
Brief Title: High Energy Density Pulse Electromagnetic Field for Patients With Adhensive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Liang-Cheng Chen, Director, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C202305036
Record Dates: First submitted 2023-08-12; First posted 2023-08-21 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Adhesive Capsulitis
Keywords: adhesive capsulitis; high energy density pulse electromagnetic field
MeSH Terms: conditions — Bursitis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physiotherapy and high-PEMF (Experimental): The patient receives physiotherapy and high-PEMF therapy twice weekly, over a period of three weeks.
  Interventions: Device: High energy density pulse electromagnetic field; Other: physiotherapy
- physiotherapy and sham high-PEMF (Sham Comparator): The patient receives physiotherapy and sham high-PEMF therapy twice weekly, over a period of three weeks.
  Interventions: Other: physiotherapy; Device: sham High energy density pulse electromagnetic field

INTERVENTIONS:
Device: High energy density pulse electromagnetic field — The treatment coil is positioned over the area of the shoulder that experiences the most pain, and it remains in place for a duration of 9 minutes. The patient is subjected to a high-energy high-PEMF with a frequency of 3 pulses per second during the session.
  Arms: physiotherapy and high-PEMF
Other: physiotherapy — Physiotherapy includes a range of activities such as passive and active-assisted shoulder range of motion (ROM) exercises, Pendulum exercises, Codman's exercises, and Cross-body reach exercises. These exercises are conducted under the supervision of a physiotherapist and each training session lasts approximately 30 minutes.
Device: sham High energy density pulse electromagnetic field — The sham treatment coil is positioned over the area of the shoulder where maximum pain is experienced, and it remains in place for a duration of 9 minutes. The parameters are consistent with those used in the experimental group. The key distinction lies in the fact that the energy output is not delivered to the patient.
  Arms: physiotherapy and sham high-PEMF

SUMMARY:
The aim of our study is to investigate the efficacy of high energy density pulse electromagnetic field for patients with adhesive capsulitis

DETAILED DESCRIPTION:
Adhesive capsulitis, a condition causing shoulder pain and limited range of motion (ROM), is estimated to affect 2-5% of the general population. Typically occurring in middle-aged individuals during their 50s to 70s, it presents with gradually developing shoulder pain and restricted ROM, particularly in external rotation.

In cases of primary adhesive capsulitis, the condition often resolves on its own, lasting around 18-24 months. However, some individuals experience persistent symptoms beyond 3 years, with up to 40% of patients and 15% facing lasting disability. Therefore, effective treatment is essential to alleviate the pain and disability associated with frozen shoulder.

High energy density pulse electromagnetic field (High-PEMF) differs from traditional PEMF and possesses the following characteristics:

Brief pulse duration (50μs) with a damped oscillation. Wide bandwidth (200kHz~300MHz) centered around 240kHz. High voltages (up to 40 kV) and peak currents (up to 10 kA) in the applicator spool.

Delivery of around 96Ws (Joule) of energy per pulse with a magnetic flux density of 50~100mT.

Tissue and organ penetration up to 20 cm. Although High-PEMF has shown positive results in chronic tendinopathy, there is limited evidence of its effectiveness in treating adhesive capsulitis. Therefore, our study aims to explore the efficacy and potential mechanisms underlying the use of High-PEMF in treating adhesive capsulitis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Physicians diagnose frozen shoulder by considering the patient's medical background, conducting a physical assessment, and reviewing X-ray and ultrasound findings.
2. The symptoms endure for a duration exceeding 3 months.
3. There exists a decrease of no less than 30 degrees in a minimum of two joint angles of the affected shoulder, namely flexion, abduction, and external rotation, in comparison to the corresponding angles of the unaffected side.

Exclusion Criteria:

1. Musculoskeletal ultrasound of the shoulder identifies a full-thickness tear or substantial tear in the rotator cuff tendons or presents calcific tendinitis.
2. Presence of systemic rheumatic disease.
3. Prior history of shoulder fracture or surgical intervention involving the shoulder joint.
4. Acute compression of cervical nerve root.
5. Patients displaying instability (e.g., those with signs of internal bleeding) or individuals with cancer.
6. Recent receipt of shoulder injections for treatment within the last 3 months.
7. Impaired cognitive function that hinders the patient's ability to provide informed consent or engage in rehabilitation therapy.
8. Expectant or breastfeeding women.
9. Meets any of the contraindications for high-energy electromagnetic pulse therapy: individuals with organ transplants, implanted cardiac pacemakers, defibrillators, metal implants (such as stents), cochlear implants, and those requiring insulin supplementation.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in pain Visual Analogue Scale(VAS) | the change from baseline, post-intervention immediately, post-intervention 1, 3, 6 months
  The visual analogue scale (VAS) is a scale used to determine the pain intensity experienced by individuals. "0" means painless and "10" means extremely painful.

SECONDARY OUTCOMES:
Change in Shoulder Pain and Disability Index (SPADI) | the change from baseline, post-intervention immediately, post-intervention 1, 3, 6 months
  Shoulder functionality and impairment were assessed employing the Chinese version of the Shoulder Pain and Disability Index (SPADI). This self-reported questionnaire comprises distinct pain and disability sections, yielding both domain-specific and overall scores. The SPADI encompasses five pain-related inquiries and eight disability-related questions, all pertaining to various shoulder issues encountered within the preceding week. Each item's score ranges between 0 (indicating no pain/normalcy) and 10 (reflecting maximal pain/impairment). The cumulative pain score ranges from 0 to 50, while the disability score ranges from 0 to 80. A higher score indicates a greater level of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Liang cheng Chen, MD, MS, Principal Investigator — Department of Physical Medicine and Rehabilitation, Tri-Service General
Locations (1):
- Tri-service general hospital, Taipei, Taiwan